CLINICAL TRIAL: NCT03880929
Title: Epidemiologic Features of Kawasaki Disease in Shanghai From 2013 Through 2017
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Children's Hospital (Other); Shanghai Children's Medical Center (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: KD EP4
Record Dates: First submitted 2019-03-06; First posted 2019-03-19 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Mucocutaneous Lymph Node Syndrome
Keywords: kawasaki disease; coronary artery lesion; epidemiology
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
To investigate the epidemiologic features of Kawasaki disease (KD) in Shanghai from 2013 through 2017 and identify the risk factors for coronary artery lesions.

DETAILED DESCRIPTION:
Based on the KD research group network established during the first survey in Shanghai, a set of questionnaires and diagnostic guidelines for KD will be sent to 50 hospitals providing pediatric medical care in Shanghai, China. Medical records of participants with KD diagnosed from January 2013 through December 2017 will be retrospectively analyzed. Data are collected by pediatricians, including demographic information, clinical manifestations, prognosis, laboratory indexes, treatment and echocardiographic findings.

Age and seasonal distribution at onset, treatment and cardiac abnormalities wil be described. Univariate and multivariate analyses will be performed to identify risk factors for coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

- meeting the diagnostic criteria for Kawasaki disease released by American Heart Association 2017

Exclusion Criteria:

* not in acute phase;
* repeated cases;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All hospitalized patients diagnosed with Kawasaki disease in Shanghai from 2013 through 2017
Sampling Method: Non-Probability Sample
Enrollment: 4533 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of coronary artery lesions | from admission to one month after onset
  Coronary artery lesions were identified with two-dimensional echocardiography in the acute phase (within one month of onset). Participants were considered to have coronary artery lesions if the luminal diameter of a coronary artery was >3.0 mm in children aged younger than 5 years or >4.0 mm in those aged 5 years and older, or when the internal diameter of a segment was ≥1.5 times that of an adjacent segment.

SECONDARY OUTCOMES:
Incidence of intravenous immunoglobulin resistance | from admission to discharge (about two weeks after onset)
  Ear temperature was measured each day during hospitalization. Intravenous immunoglobulin (IVIG) resistance was defined as persistent fever (>38°C) after 36 hours of completion of initial IVIG infusion or recurrent fever requiring another dose of IVIG or other adjunctive therapies.
Risk factors associated with coronary artery lesions | from admission to one month after onset
  Multivariate logistic regressions were performed to identify risk factors that were independently associated with coronary artery lesions. Odds ratio and 95% CI were calculated for each variable.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Liu, Dr., Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen JJ, Ma XJ, Liu F, Yan WL, Huang MR, Huang M, Huang GY; Shanghai Kawasaki Disease Research Group. Epidemiologic Features of Kawasaki Disease in Shanghai From 2008 Through 2012. Pediatr Infect Dis J. 2016 Jan;35(1):7-12. doi: 10.1097/INF.0000000000000914. PMID 26372452
- [Background] McCrindle BW, Rowley AH, Newburger JW, Burns JC, Bolger AF, Gewitz M, Baker AL, Jackson MA, Takahashi M, Shah PB, Kobayashi T, Wu MH, Saji TT, Pahl E; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee of the Council on Cardiovascular Disease in the Young; Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Surgery and Anesthesia; and Council on Epidemiology and Prevention. Diagnosis, Treatment, and Long-Term Management of Kawasaki Disease: A Scientific Statement for Health Professionals From the American Heart Association. Circulation. 2017 Apr 25;135(17):e927-e999. doi: 10.1161/CIR.0000000000000484. Epub 2017 Mar 29. PMID 28356445
- [Background] JCS Joint Working Group. Guidelines for diagnosis and management of cardiovascular sequelae in Kawasaki disease (JCS 2008)--digest version. Circ J. 2010 Sep;74(9):1989-2020. doi: 10.1253/circj.cj-10-74-0903. Epub 2010 Aug 18. No abstract available. PMID 20724794

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT03880929/Prot_SAP_000.pdf